CLINICAL TRIAL: NCT07392125
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Phase 3 Trial Evaluating the Efficacy and Safety of Cytisinicline for Vaping Cessation in Adults Using Nicotine-Containing E Cigarettes
Brief Title: Phase 3 Trial Evaluating the Efficacy and Safety of Cytisinicline for Vaping Cessation in Adults Using Nicotine-Containing E Cigarettes
Acronym: ORCA-V2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-CYT-12
Record Dates: First submitted 2026-01-20; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Vaping Cessation
Keywords: vaping cessation
MeSH Terms: interventions — cytisine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Placebo Comparator): 12 weeks of placebo + behavioral support; 400 subjects
  Interventions: Drug: Placebo; Behavioral: Behavioral Support
- Arm B (Active Comparator): 12 weeks cytisinicline + behavioral support; 400 subjects
  Interventions: Drug: Cytisinicline; Behavioral: Behavioral Support

INTERVENTIONS:
Drug: Cytisinicline — Tablet, 3 times a day (TID), 12 weeks
  Other Names: cytisine
  Arms: Arm B
Drug: Placebo — Tablet, 3 times a day (TID), 12 weeks
  Arms: Arm A
Behavioral: Behavioral Support — 16 behavioral support sessions, starting prior to randomization and through Week 12, 3 additional sessions during the follow-up period.

SUMMARY:
This will be a multi-center, double-blind, randomized, placebo-controlled, Phase 3 study conducted in male or female adults who are daily nicotine e-cigarette users only.

A total of approximately 800 subjects will be randomly assigned (1:1) to one of two Arms:

* Arm B, 12 weeks cytisinicline + behavior support: N=400 or
* Arm A, 12 weeks of placebo+ behavior support: N=400) The primary objective is to assess whether subjects randomized to Arm B (3 mg cytisinicline TID for 12 weeks plus behavioral support) have a higher probability of nicotine vaping cessation from Week 9 to Week 12 as compared to subjects randomized to Arm A (placebo TID for 12 weeks plus behavioral support).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age ≥18 years.
* Test positive for cotinine using a point-of-care Oral Fluid Screening Device (OFD) with positive detection at ≥30 ng/mL cotinine.
* Current daily nicotine-containing electronic cigarette usage as recorded in a screening diary for at least 7 consecutive days. Willing to bring the e-cigarette or nicotine device used to the clinical site so that the specific product type, flavor, and nicotine level can be documented.
* Failed at least one previous attempt to stop vaping with or without therapeutic support.
* Willing to initiate study treatment on the day after randomization and set a quit date within Day 7 and Day 14.
* Willing to actively participate in the study's vaping cessation behavioral support provided throughout the study.
* Able to fully understand study requirements, willing to participate, and comply with dosing schedule.
* Sign the Informed Consent Form.

Exclusion Criteria:

* Currently smoking or having smoked within 3 months prior to study randomization, any combustible cigarettes, other combustible tobacco products or non-combustible tobacco products such as heat not burn products or nicotine pouches (ie, dual users).
* Currently smoking/vaping cannabis or having smoked or vaped cannabis within 4 weeks (28 days) prior to study randomization or planned use while on study. Other methods of cannabis consumption, eg, edibles, tinctures, capsules, topicals, etc. are allowed.
* Expired Carbon Monoxide (CO) levels ≥6 ppm, indicating recent combustible tobacco or cannabis smoking.
* A score of 0-3 on the Penn State e-Cigarette Dependence Index indicating no dependence.
* More than 1 study subject in same household during the study treatment period.
* Known hypersensitivity to any of the excipients, previous cytisinicline treatment in a prior clinical study, or any previous use of cytisinicline.
* Positive urinary drugs of abuse screen determined within 28 days before the first dose of study drug. (Note: Although THC is part of the standard drug screen, it is not necessarily exclusionary. Refer to exclusion criteria #2).
* Clinically significant abnormal serum chemistry or hematology values, as determined by the investigator, within 28 days of randomization.
* Clinically significant abnormalities on screening visit 12-lead ECG, as determined by the investigator, after minimum of 5 minutes in supine position within 28 days of randomization.
* Recent history (within 3 months prior to screening) of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident or hospitalization for congestive heart failure.
* Current uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg).
* Currently psychotic or having had a psychotic event in the 3 months prior to the screening visit. If any subject becomes psychotic during the study, they must be removed from treatment and/or additional study visits.
* Currently having suicidal ideation or risk for suicide (YES to either question 3, 4 or 5 OR YES to any suicidal behavior question on the C-SSRS with clear suicidal intent or suicide attempt within the last 10 years).
* Current symptoms of moderate to severe depression (depression score ≥11 using depression questions on the Hospital Anxiety and Depression Scale [HADS] at screening visit).
* Renal impairment defined as a creatinine clearance (CrCl) <60 mL/min at screening visit (estimated with the Cockroft-Gault equation and reported by the central laboratory).
* Hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0 x the upper limit of normal (ULN) at screening visit.
* Recent history or symptoms (within 4 weeks of randomization) of unstable respiratory disease (eg, pneumonia, product-use associated lung injury or EVALI, etc).
* Women who are pregnant or breast-feeding.
* Female subjects of childbearing potential who do not agree to use acceptable methods of birth control during the study. Acceptable methods of birth control include:
* True abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
* Barrier methods:
* diaphragm
* cervical cap
* contraceptive sponge
* intrauterine device (IUD)
* double barrier method (condom with spermicide)
* Hormonal methods:
* Oral contraceptives
* Vaginal ring such as NuvaRing
* Skin patch such as Xulane
* Injection such as Depro-Provera
* Implantable rod such as Nexplanon
* Intrauterine device (IUD)
* Participation in a clinical study with an investigational drug or biologic in the 4 weeks prior to study randomization.
* Use of any smoking cessation medications (bupropion, varenicline, nortriptyline, or any nicotine replacement therapy [NRT]) in the 4 weeks prior to study randomization or planned use of these or other nicotine replacement medications during the study.
* Any planned use during the study of combustible cigarettes or other nicotine-containing, non-vaping products (eg, pipe tobacco, cigars, snuff, smokeless tobacco, hookah, ZYN pouches, etc).
* Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Objective | Randomization to Week 24 follow-up visit
  Assess whether subjects randomized to Arm B (3 mg cytisinicline TID for 12 weeks plus behavioral support) have a higher probability of nicotine vaping cessation from Week 9 to Week 12 post-randomization as compared to subjects randomized to Arm A (placebo TID for 12 weeks plus behavioral support). Successful vaping cessation is defined as weekly vaping abstinence during the last 4 weeks of the 12-week treatment period (Week 9 through Week 12) using quantitative cotinine levels at <10 ng/mL for biochemical verification and subject's self-report of no vaping using a daily electronic diary

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ball, Study Director — Achieve Life Sciences, Inc.